CLINICAL TRIAL: NCT05638789
Title: Endoscopic Sphincterotomy With Balloon Dilatation Versus Sphincterotomy Alone For Common Bile Duct Stones Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, OOI JIE SOANG, PRINCIPAL INVESTIGATOR, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUSM
Record Dates: First submitted 2022-10-24; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Choledocholithiasis
Keywords: endoscopic sphincterotomy (EST); endoscopic papillary large balloon dilatation (EPLBD)
MeSH Terms: conditions — Choledocholithiasis | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Intervention Model Description: EST alone versus EST + EPLBD group
Who Masked: Participant
Masking Description: 66 patients with CBD stone will be divided into two groups which is Group A(EST+EPLBD) (33 cases) and Group B (EST alone) (33 cases). Randomization will be done using computer software for sequence generation and was stratified with 1:1 allocation using random block sizes of 6 and 8 to Group A or Group B. The allocation concealment mechanism was developed by preparing 88 sealed and opaque envelopes. Each envelop contain one allocation sequence which is generated by computer software. Data collection officer will randomly open one of the envelop each time one patient recruited and will need to follow the allocation sequences inside the envelop in order to determine whether the patient to be Group A or Group B patient. This is single blinded study whereby the participant is blinded but the endoscopist is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EST alone (Active Comparator)
  Interventions: Procedure: endoscopic sphincterotomy (EST) versus EST plus endoscopic papillary large balloon dilatation (EPLBD)
- EST + EPLBD (Active Comparator)
  Interventions: Procedure: endoscopic sphincterotomy (EST) versus EST plus endoscopic papillary large balloon dilatation (EPLBD)

INTERVENTIONS:
Procedure: endoscopic sphincterotomy (EST) versus EST plus endoscopic papillary large balloon dilatation (EPLBD) — EST alone vs EST plus EPLBD in removing common bile duct stone

SUMMARY:
Gallstone is a worldwide clinical problem which affecting most of the populations with incidence of 15 to 20% in west and 10% in Asians. About 5 to 15% of patient with gallstone will go on to develop bile duct calculi. There are several endoscopic strategies developed for treatment of common bile duct stone such as endoscopic sphincterotomy (EST), endoscopic papillary large balloon dilatation (EPLBD) and combination of EST plus EPLBD. Our aim of this study is to compare efficacy, and safety of EST alone group versus EST plus EPLBD group in removing CBD stone.

DETAILED DESCRIPTION:
Endoscopic sphincterotomy (EST) is most widely used during endoscopic retrograde cholangiopancreatography (ERCP) to remove common bile duct (CBD) stone and considered as standard therapy for treatment of choledocholithiasis. However, in view of EST requires an adequate incision on major duodenal papilla to achieve biliary cannulation, it can potentially cause damage to biliary sphincter during the procedure and potentially increased risk of some complications such as bleeding and biliary reflux. This procedure carries risk of complications such as haemorrhage, perforation, and long-term effect like sphincter dysfunction.

Staritz introduced a method called endoscopic papillary large balloon dilatation (EPLBD) in 1983 as an alternative to EST in clearing CBD stone. EPLBD can reduced the risk of bleeding and perforation post procedure, but it carries higher risk of post-ERCP pancreatitis.

About 10 to 15% of CBD stone are unable to be extracted by both EST or EPLBD alone, especially in those patients with big and difficult stone (size bigger than 10 to 15mm, numerous, barrel-shaped, and impacted stones). Besides that, other factors that can contribute to failure of stone extraction are periampullary diverticulum or post operative variation, tortuosity and tightening of distal common bile duct.

In 2003, Ersoz introduced combination of EST plus EPLBD as an alternative method. It can reduce the risk of complications through avoiding a complete sphincterotomy, shortening procedural time, and reducing the need of usage of mechanical lithotripsy.

In a study on 2007, it showed that EST plus EPLBD had comparable efficacy and safety when compared to conventional EST alone and both groups have similar complication rate. Besides that, in a recent study in 2020, it also showed that EST plus EPLBD had a comparable efficacy when compared with EST alone in clearing CBD stone and EST plus EPLBD required shorter procedural time when compared with EST alone. There is no significant increased risk in pancreatitis for EST plus EPLBD. While, in a randomized controlled study in 2017, it showed that EST plus EPLBD is more effective than EST alone in clearing large CBD stone and is equally safe compared to EST alone. In another randomized controlled trial in 2013, the study showed that the success rate for complete CBD stone removal in first session is higher in EST plus EPLBD group when compared to EST alone and it is statistically significant. But the overall stone clearance rate and complication rate was similar in both groups. Apart from that, there are many other studies have suggested EST plus EPBD as a safe and promising alternative to conventional EST or EPLBD. In a published meta-analysis, accumulated data showed that EST plus EPLBD is a safe and effective procedure in removing large or difficult CBD stone without any additional risk of complications.

There is still no definite conclusion in evaluating superiority of EST plus EPLBD vs EST alone in term of efficacy in removing CBD stone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age 18 and above
2. Patient with CBD stone documented on imaging studies

Exclusion Criteria:

1. CBD stone size more than 15mm
2. CBD stone number more than 3
3. Concurrent hepatobiliary tumour
4. Intrahepatic stone
5. Bleeding tendencies: coagulopathy, thrombocytopenia, patient on anticoagulant medication
6. Patient in sepsis/ Cholangitis patient
7. Patient with acute pancreatitis
8. Prior history of Bilroth II or Roux-en-y surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Rate of complete common bile stone clearance of EST alone versus EST plus EPLBD | 12 months
  to compare the rate of overall complete stone clearance in EST alone arm vs EST plus EPLBD arm
Complication rate of EST alone versus EST plus EPLBD in removing CBD stone | 12 months
  to compare complication rate which are post ERCP bleeding, post-ERCP pancreatitis, perforation and cholangitis rate of EST alone arm versus EST plus EPLBD arm in removing CBD stone

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery School of Medical Sciences, Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Result] Suissa A, Yassin K, Lavy A, Lachter J, Chermech I, Karban A, Tamir A, Eliakim R. Outcome and early complications of ERCP: a prospective single center study. Hepatogastroenterology. 2005 Mar-Apr;52(62):352-5. PMID 15816433
- [Result] Staritz M, Ewe K, Goerg K, Meyer zum Buschenfelde KH. Endoscopic balloon tamponade for conservative management of severe hemorrhage following endoscopic sphincterotomy. Z Gastroenterol. 1984 Nov;22(11):644-6. PMID 6516498
- [Result] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Result] Fu BQ, Xu YP, Tao LS, Yao J, Zhou CS. Endoscopic papillary balloon intermittent dilatation and endoscopic sphincterotomy for bile duct stones. World J Gastroenterol. 2013 Apr 21;19(15):2425-32. doi: 10.3748/wjg.v19.i15.2425. PMID 23613639
- [Result] Shim CS, Kim JW, Lee TY, Cheon YK. Is endoscopic papillary large balloon dilation safe for treating large CBD stones? Saudi J Gastroenterol. 2016 Jul-Aug;22(4):251-9. doi: 10.4103/1319-3767.187599. PMID 27488319
- [Result] Attam R, Freeman ML. Endoscopic papillary large balloon dilation for large common bile duct stones. J Hepatobiliary Pancreat Surg. 2009;16(5):618-23. doi: 10.1007/s00534-009-0134-2. Epub 2009 Jun 24. PMID 19551331